CLINICAL TRIAL: NCT04037488
Title: Body Compositions Change in Patients With Prostate Cancer Treated With Androgen Deprivation Therapy
Brief Title: Changes in Body Composition With Patients Under Androgen Deprivation Therapy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Seoul National University Hospital (Other)
Collaborators: HanAll BioPharma Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: SNUH-URO-2018-01
Record Dates: First submitted 2018-11-29; First posted 2019-07-30 (Actual); Last update posted 2019-07-30 (Actual); Status verified 2018-09

CONDITIONS: Sarcopenia; Prostate Cancer
Keywords: Androgen deprivation therapy; Prostate cancer; Body composition; Lean body mass
MeSH Terms: conditions — Sarcopenia; Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Cohort: ADT patients: All enrolled patient data entered in single group cohort. All patient who started androgen deprivation therapy for prostate cancer can included this cohort by following inclusion and exclusion criteria. We do not planned any intervention on this cohort. We measuring changes of body composition by Inbody 320 in the planned follow-up period.
  We planned sub-group analysis for timing of intervention (Intervention 1) , ADT type(Intervention 2), LHRH agonist type(Intervention 3), patients age(Intervention 4), initial PSA level (Intervention 5) and Gleason Grade Group (Intervention 6).
  Interventions: Diagnostic Test: Inbody 320

INTERVENTIONS:
Diagnostic Test: Inbody 320 — Total Skeletal muscle mass (SMM), Skeletal muscle index (SMI), Relative Skeletal muscle mass index (RASM), Fat body mass (FBM), Body mass index (BMI), Body fat percentage, Body water content, Edema Value were calculated by Inbody 320
  Other Names: Body composition change

SUMMARY:
This study aimed to evaluate the correlation of change in body composition and oncological outcomes of prostate cancer patients under androgen deprivation therapy(ADT).

DETAILED DESCRIPTION:
Sarcopenia, decrease lean body mass (LBM) is the well-known parameter which negatively related to physical activity, morbidity and patients survival. Aging and decreased blood androgen level are well known risk factors of sarcopenia in male population.

Androgen deprivation therapy (ADT) is commonly performed in advanced or recurred prostate cancer patient and lead to accelerating decreasing blood androgen level. The previous studies defined the sarcopenia after ADT by calculated the (muscle component area) / (total body area) on computed tomography (CT) scan. However, CT scan is not recommended for routine follow up examination of ADT patients thus this measurement of sarcopenia has limitation on clinical usage.

This study using Inbody 320 for measure body composition. Inbody 320 based on multi-frequency Bioelectrical Impedance Analysis(BIA) method that calculated specific body component by differences in impedance indexes of fat, muscle and extracellular body fluid. Inbody measurement show precision accuracy and safety on body composition measurement, thus it frequently used in studies of obesity, nutrition and sports fields.

We calculating the total skeletal muscle mass (SMM), skeletal muscle index(SMI), relative skeletal muscle mass index (RASM), fat body mass (FBM), body mass index (BMI), body fat percentage, body water content, and edema value by Inbody 320 in the patients who treated by ADT in prostate cancer patients. Enrolled patients check the body composition parameters at the baseline (before ADT) and after ADT 3,6,12,18,24 months.

We prospectively measuring the 2 years changes of body composition and sarcopenia after ADT treatment. Patients characteristics (Age, underlying disease), Prostate cancer status (PSA level, Gleason grade group, initial treatment), ADT methods characters (timing, type) and oncological outcome (Recurrence, Metastasis, Castration resistance) were measuring in the cohort population.

Post hoc analysis were performed in the timing (initial, salvage or adjuvant) or type (LHRH agonist, Antiandrogen or surgical castration) of ADT for development of sarcopenia. Sub-arm analysis were performed for assessing that effect of presence of sarcopenia on oncological outcome and functional outcomes after ADT.

ELIGIBILITY:
Inclusion Criteria:

* Age over 20 year-old
* Patient with ECOG-PS 0 to 2
* Prostate cancer patients
* Considered Androgen deprivation therapy with any cause
* Patient agreed with informed consent of this study

Exclusion Criteria:

* History of previous ADT
* Planned intermittent treatment or short term ADT (less than 2 year)
* Contraindication of ADT
* Severe cognitive impairment, who cannot eligible for survey
* Secondary malignancy
* Patient cannot perform InBody test because of physical or underlying disease.

Min Age: 20 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with long-term (more than 2 year) androgen deprivation therapy for treatment of prostate cancer, without any other malignancy.
Sampling Method: Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2019-08 (Estimated); Primary Completion 2021-10-30 (Estimated); Study Completion 2021-10-30 (Estimated)

PRIMARY OUTCOMES:
Body composition change-Skeletal muscle index (SMI) | Baseline (preADT) and Post ADT 3, 6, 12, 18, 24 months
  Lean body mas (kg) / body weight (kg) x 100 (%)
Body composition change-Body mass index (BMI) | Baseline (preADT) and Post ADT 3, 6, 12, 18, 24 months
  {body weight (kg)} / {height (m)^2}
Body composition change-Relative skeletal muscle index (RASM) | Baseline (preADT) and Post ADT 3, 6, 12, 18, 24 months
  Sum of skeletal muscle mass in limbs (kg) / {height (m)^2}
Body composition change - fat body mass (FBM) | Baseline (preADT) and Post ADT 3, 6, 12, 18, 24 months
  fat body mass (FBM) calculated by Inbody 320

SECONDARY OUTCOMES:
Laboratory changes-PSA | Baseline (preADT) and Post ADT 3, 6, 12, 18, 24 months
  PSA level changes
Laboratory changes-Testosterone | Baseline (preADT) and Post ADT 3, 6, 12, 18, 24 months
  Testosterone level changes
Oncologic outcomes - recurrence | Up to 24 weeks
  Any local or distance recurrence
Oncologic outcomes - survival | Up to 24 weeks
  Any cause of death

CONTACTS AND LOCATIONS:
Overall Officials: Chang Wook Jeong, MD. PHD., Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea